CLINICAL TRIAL: NCT01262339
Title: Randomized, Single-blind Comparison of Botulinum Toxin Treatment for Palmar Hyperhidrosis Via Iontophoresis Versus Intradermal Injection
Brief Title: BTX-A Treatment for Palmar Hyperhidrosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low enrollment; principal investigator left sponsoring institution
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Allergan (Industry); Mattioli (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-2009-0193
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Primary Focal Hyperhidrosis of the Hands
Keywords: Primary focal hyperhidrosis; interdermal injections; iontophoresis; BTX-A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Comparator of Hand A intervention vs Hand B (Active Comparator): Hand A will receive 100U of BTX-A injected intradermally (SOC) Hand B will receive 100U delivered via iontophoresis.
  Interventions: Drug: BTX-A

INTERVENTIONS:
Drug: BTX-A — 100 units of BTX-A will be delivered subject's hand via iontophoresis and standard of care intradermal injection of 100 units BTX-A will be delivered to the contra-lateral hand
  Other Names: botulinum Toxin A

SUMMARY:
Primary focal hyperhidrosis (excessive sweating) is a debilitating condition affecting approximately 3% of the population in the United States. Not only that it is a major social embarrassment to affected individuals, it also has significant negative impacts on career, school, and relationship. Botulinum toxin A (BTX-A), a sterile neurotoxin purified from Clostridium bacteria, was approved by the U.S. Food & Drug Administration in 2004 for the treatment of severe focal axillary hyperhidrosis that does not respond to topical antiperspirants. It is becoming a promising treatment for many patients suffering this condition. Over the past decade, the medication has also been used effectively for many other forms of focal hyperhidrosis such as the hands, feet, forehead, scalp and groin. Unfortunately, BTX-A injection for primary focal hyperhidrosis of the palms and soles are often limited by pain and post treatment muscle weakness associated with the procedure. Recent studies have demonstrated that BTX-A can be delivered across the skin via electric current using a medical device, called iontophoresis (FDA 510(k) clearance # K042590 or Phoresor IIPM700). Studies with limited number of patients have demonstrated promising results with this new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female
* Age 16 and older
* If <18, parent/legal guardian willing to sign consent and accompany to visits
* Diagnosis of hyperhidrosis disease with a severity score (HDSS) of 3 or 4
* Treatment types of topical antiperspirants, iontophoresis, or systemic anticholinergics have failed to treat
* Able to come to 5 clinical visits during the study period

Exclusion Criteria:

* Diagnosis of neuromuscular disease such as peripheral motor neuropathic diseases (e.g. amyotrophic lateral sclerosis, or motor neuropathy)
* Diagnosis of neuromuscular junctional disorders (e.g. myasthenia gravis or Lambert-Eaton syndrome)
* Diagnosis of dysphagia
* Individuals with surgical implants such as pacemakers, orthopedic hardware, etc.
* Individuals who are Immunocompromised
* Systemic infectious illness or infection at the injection site(s)
* Known hypersensitivity to any ingredient in the formulation of the drug
* Organic cause of hyperhidrosis
* Known allergy to the ingredients in the general anesthesia
* Diagnosis of cardiac/pulmonary issues or disease
* Women who are pregnant or suspected to be pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comparator of Hand A Intervention vs Hand B
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Comparator of Hand A Intervention vs Hand B
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Efficacy of Botulinum Toxin A (BTX-A) in the Treatment of Primary Palmar Hyperhidrosis Delivered Via Iontophoresis.
Time Frame: 26 weeks
Population: Study was closed prematurely as principal investigator left the University of Wisconsin. Insufficient data for outcome measures analysis. Data was not entered into tabular format. Study closed and records archived.
Groups:
- Active Comparator: Comparator of Hand A Intervention vs Hand B: Hand A will receive 100U of BTX-A injected intradermally (SOC) Hand B will receive 100U delivered via iontophoresis.
Arm/Group | Active Comparator: Comparator of Hand A Intervention vs Hand B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Comparator of Hand A Intervention vs Hand B
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No